CLINICAL TRIAL: NCT04054843
Title: Afamin Levels in First Trimester Pregnancies With Gestational Diabetes Mellitus
Brief Title: Afamin in Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Aykan Yucel, Professor, M.D., Professor, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Other Study IDs: Afamin in GDM
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gestational diabetes mellitus: First trimester pregnancies with gestational diabetes mellitus
  Interventions: Diagnostic Test: Afamin
- Control: First trimester healthy pregnancies
  Interventions: Diagnostic Test: Afamin

INTERVENTIONS:
Diagnostic Test: Afamin — Plasma maternal afamin levels

SUMMARY:
This study includes pregnancies in 11 to 14 th gestational weeks. Investigators will sample maternal plasma in the first trimester and analyze maternal plasma afamin values. All these women will then be screened by two step OGTT. Investigators will compare afamin levels in GDM and control groups.

DETAILED DESCRIPTION:
Background Gestational diabetes mellitus (GDM) is an endocrinopathy that occurs during pregnancy, and presents several clinical findings together with increased blood glucose levels. The frequency of GDM differs, while the incidence of the disease in Turkey is reported to be 7%. Most of the societies recommend screening all women with or without any risk factors in terms of GDM. The definitive diagnosis is made via oral glucose challenge test (OGTT). Early diagnosis and treatment are the key points to improve maternal and fetal outcomes. Different biomarkers are studied regarding GDM diagnosis starting from first trimester. However, there is not a worldwide accepted biomarker for defining the high risk group to the date. Afamin is known as an important indicator of oxidative stress. Moreover, oxidative stress itself is strongly associated with insulin resistance and obesity which are responsible from GDM pathogenesis.

Objective To investigate the association between first trimester maternal plasma afamin levels and GDM. Also, investigators aimed to understand the role of afamin for the prediction of GDM in this study.

Methods This is an observational prospective cohort study conducted in Department of Perinatology, Etlik Zubeyde Hanim Women's Health Care, Training and Research Hospital, University of Health Sciences, Ankara, Turkey. During 11 and 14 weeks of gestational, maternal blood will be obtained from eligible pregnant women, and samples will be stored at -80 oC. Informed written consent will be obtained from participants. Between 24th and 28th gestational weeks, all these women will be screened by two step OGTT. Then, afamin levels will be compared in GDM and control groups. Exclusion criteria are; multiple pregnancy, fetal anomalies, pregestational diabetes, underlying chronic diseases (hypertension, thyroid dysfunction, other endocrinopathies, autoimmune disorders), age <18 or > 35 years, fasting glucose level > 105 mg/dL or random glucose level > 200 mg/dL.

ELIGIBILITY:
Inclusion criteria:

* singleton pregnancy,
* having no fetal anomalies
* having no pregestational diabetes
* having no underlying chronic diseases (hypertension, thyroid dysfunction, other endocrinopathies, autoimmune disorders)
* age >18 or < 35 years
* fasting glucose level < 105 mg/dL

Exclusion Criteria:

* multiple pregnancy
* fetal anomalies
* pregestational diabetes
* underlying chronic diseases (hypertension, thyroid dysfunction, other endocrinopathies, autoimmune disorders)
* age <18 or > 35 years
* fasting glucose level > 105 mg/dL or random glucose level > 200 mg/dL

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Women within 11 and 14 weeks of gestational weeks
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Maternal plasma afamin levels In first trimester GDM prediction | 6 months
  The predictive value of first trimester maternal plasma afamin levels for the diagnosis of gestational diabetes mellitus in comparison with two step OGTT

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided